CLINICAL TRIAL: NCT05103514
Title: The Longitudinal Impact of Socioeconomic Status and the Competing Neurobehavioral Decision Systems on Recovery From Substance Use Disorder
Brief Title: The Longitudinal Impact of SES and the CNDS on Recovery From SUD
Status: Not yet recruiting | Type: Observational
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Jeffrey Stein, Professor, Virginia Polytechnic Institute and State University
Other Study IDs: SES- Longitudinal Study
Record Dates: First submitted 2021-10-07; First posted 2021-11-02 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1: Participants in this group started their recovery process < 1 year ago
  Interventions: Other: Online Survey
- Cohort 2: Participants in this group started their recovery process 1 to <2 years ago
  Interventions: Other: Online Survey
- Cohort 3: Participants in this group started their recovery process 2 to <3 years ago
  Interventions: Other: Online Survey

INTERVENTIONS:
Other: Online Survey — There are no interventions planned for this study. This is an observational study only.

SUMMARY:
The goal of this study is to provide a scientific understanding of the impact of socioeconomic status (SES) on the recovery trajectory (psychosocial functioning, relapse/remission status, and neurocognitive mechanisms).

DETAILED DESCRIPTION:
The study will characterize the effect of SES (subjective and objective indicators) on long-term trajectories of recovery and neurocognitive functioning. By using an accelerated longitudinal design, the investigators will examine the association between baseline SES, changes in CNDS, and changes in psychosocial functioning (e.g., quality of life) and relapse. Moreover, the investigators will use computational modeling to capture underlying changes in components of CNDS functioning related to SES and SUD recovery.

ELIGIBILITY:
Inclusion Criteria:

1. be ≥18 yrs old
2. meet lifetime DSM-5 SUD criteria
3. have a Recovery Initiation Date less than 3 years prior to the time of enrollment
4. be able to read independently
5. be free of legal problems that could limit participation
6. reside in the U.S.
7. anticipate continued Internet access (to ensure ongoing contact and data collection)
8. be a registrant of the International Quit and Recovery Registry (IQRR)

Exclusion Criteria:

1. Minors will not be included
2. Prisoners will not be included. If participants become incarcerated during this study, they will not be contacted to complete assessments during their incarceration. If the incarceration ends during the study, they may be contacted to participate in assessments.
3. Adults who are not capable of consenting on their own behalf

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals in recovery from SUD who meets the study inclusion criteria will be recruited from The International Quit & Recovery Registry (IQRR) (https://quitandrecovery.org). Participants will be recruited from existing or new IQRR registrants; that is, IQRR registrants meeting the inclusion criteria (see above) will be invited to participate. Also, the recruitment of new registrants will use methods designed to reflect the heterogeneity of the recovery population.
Sampling Method: Non-Probability Sample
Enrollment: 675 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in Socioeconomic Status (SES)- Individual Subjective SES | Approximately every 3 months from date of baseline session through study completion, an average of 3 years
  Individual Subjective SES will be determined using the MacArthur Scale of subjective social status. Participants will be presented with two social ladders that have 10 steps each and asked to place themselves on the rung that best represent where they stand at this time in their life (1=lowest rung and 10= highest rung), relative to other people in (1) the United States and (2) their community. Higher scores on the 10-rung ladder indicate higher subjective SES.
Change in Socioeconomic Status (SES)- Individual Objective SES | Approximately every 3 months from date of baseline session through study completion, an average of 3 years
  Individual Objective SES will be measured using a composite that was developed by the US Department of Justice (i.e. National Crime Victimization Survey Index 1) that incorporates four main SES elements (i.e., income, education, employment status, and housing tenure measures). Specifically, the SES composite index includes two individual level characteristics: education (possible range: 0-3) and employment in the last 6 months (possible range: 0-1); and two household level characteristics: income as a percentage of the federal poverty level (FPL; possible range: 0-3) and housing tenure (possible range: 0-1). The final SES score (possible range: 0-8) is collapsed into three levels: low (total score of 0 to less than 3), middle (total score of 3 to less than 6), and upper (total score of 6-8) SES.
Change in CNDS functioning | Approximately every 3 months from date of baseline session through study completion, an average of 3 years
  Delay Discounting (DD) task will be administered to assesses the value of delayed reinforcers. Participants make hypothetical choices between amounts of delayed and immediate money at various delays (e.g., 1 day to 25 years)
Change in Psychosocial Functioning- The Psychosocial Functioning Inventory (PFI) | Approximately every 3 months from date of baseline session through study completion, an average of 3 years
  The Psychosocial Functioning Inventory (PFI) will be used to measure social functioning. The social behavior sub-scale will be calculated from 10 items of the PFI and included items that assess the frequency of problematic social behavior and social interactions in the past 90 days. The psychosocial functioning scale yields a score ranging from 0-100, with higher scores indicating greater impairment.
Change in Psychosocial Functioning- World Health Organization (WHO)-Quality of Life | Approximately every 3 months from date of baseline session through study completion, an average of 3 years
  WHO-Quality of Life brief assessment (BREF) will be used to measure the four domains of quality of life: (1) physical health; (2) psychological (3) social relationships; and (4) environment (26 items). Each item in the WHOQOL-BREF will be scored with a 5-point Likert scale (three items are reverse scored), and these scores will be used to generate raw scores for each domain, which will be then scaled 0-100, with higher scores indicating greater quality of life.
Change in Psychosocial Functioning- Satisfaction with Life and social Functioning | Approximately every 3 months from date of baseline session through study completion, an average of 3 years
  Satisfaction with life and social functioning over the past 90 days will be assessed using 4 questions: How happy have you been (1) with life?; (2) with your living situation? and (3) with your relationships? and (4) Did you feel satisfied with leisure, social, and recreational activities? (0 = satisfied/happy; 1 = dissatisfied/unhappy)
Change in Psychosocial Functioning- Career Engagement | Approximately every 3 months from date of baseline session through study completion, an average of 3 years
  Engagement in proactive career behaviors over time (9 items). Each item in the career engagement measure will be scored with the 5-point Likert-type scale. The average scale scores will range between 1-5 with higher score indicating greater engagement.
Change in Psychosocial Functioning- Addiction Severity | Approximately every 3 months from date of baseline session through study completion, an average of 3 years
  The Addiction Severity Index (ASI) will be used to assess experiences of serious depression, serious anxiety or tension, and cognitive difficulty (i.e., trouble understanding, concentrating, or remembering) in the past 90 days. All items will be binary indicators, where 0 = employed or symptom not present and 1 = unemployed or symptom present. Items will be examined individually.
Change in Substance Use- SUD Status and Severity | Approximately every 3 months from date of baseline session through study completion, an average of 3 years
  The Diagnostic and Statistical Manual-5 (DSM-5) SUD (last year & last 3 months) will be used to assess SUD status and severity with mild, moderate, and severe sub-classifications
Change in Substance Use- Consumption | Approximately every 3 months from date of baseline session through study completion, an average of 3 years
  Timeline Follow Back-90 (TLFB-90) will be used to obtains retrospective daily estimates of substance use in the last 3 month. TLFB can generate a variety of variables that provide more precise and varied information (e.g., pattern, variability) about a person's substance use

CONTACTS AND LOCATIONS:
Overall Officials: Warren Bickel, PhD, Principal Investigator — Virginia Polytechnic Institute and State University

IPD SHARING:
Plan to Share IPD: No